CLINICAL TRIAL: NCT04818775
Title: Use of Sterile HemaClear Tourniquet Below Calf Versus Pneumatic Tourniquet at the Thigh for Ankle and Foot Surgery
Acronym: HemaClear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HemaClear
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Foot Fracture; Ankle Fractures; Ankle Injuries; Foot Injuries and Disorders
Keywords: Foot Fracture; Ankle Fractures; Ankle Injuries; Orthopaedic Devices Associated with Misadventures; Foot Injuries and Disorders
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries; Foot Injuries; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HemaClear (Experimental)
  Interventions: Device: HemaClear
- Pneumatic Tourniquet (Active Comparator)
  Interventions: Device: Pneumatic Tourniquet

INTERVENTIONS:
Device: HemaClear — HemaClear Model A
  Other Names: HemaClear Model A
  Arms: HemaClear
Device: Pneumatic Tourniquet — Pneumatic Tourniquet
  Arms: Pneumatic Tourniquet

SUMMARY:
This is a Randomized controlled trial evaluating the effects of the use of Sterile HemaClear Tourniquet Below Calf Versus Pneumatic Tourniquet at the Thigh for Ankle and Foot Surgery

The trial will randomize 60 patients into an experimental group with HemaClear or Active comparator group with Pneumatic Tourniquet.

The outcomes are: effectiveness of the tourniquet, bleeding escapes, infection, deep vein thrombosis, pain at the tourniquet site, neurologic problems related to the tourniquet

ELIGIBILITY:
Inclusion Criteria:

* Ankle and foot surgery

Exclusion Criteria:

* Infection
* Tumors
* Open fracture
* Burns
* Varicose veins
* Isquemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
infection rates | after 1 week
  infection rates
infection rates | after 3 months
  infection rates
Deep vein thrombosis | after 1 week
  Deep vein thrombosis (Clinical assessment and Doppler ultrasound)
Deep vein thrombosis | after 3 months
  Deep vein thrombosis (Clinical assessment and Doppler ultrasound)

SECONDARY OUTCOMES:
local pain | after 1 week
  local pain at the tourniquet site (Visual Analogue Scale)
local pain | after 3 months
  local pain at the tourniquet site (Visual Analogue Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Maurício P Barbosa, MD, Principal Investigator — Hospital do Coracao
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil